CLINICAL TRIAL: NCT00727662
Title: Iyengar Yoga for Breast Cancer Survivors With Persistent Fatigue
Brief Title: A Yoga and Wellness Program for Breast Cancer Survivors With Persistent Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Bower, Julienne, Assistant Professor, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01AT003682 (NIH)
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer; Fatigue
Keywords: Breast Cancer; Fatigue; Proinflammatory Cytokines; Physical functioning; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Yoga
  Interventions: Other: Iyengar Yoga
- 2 (Active Comparator): A Wellness Seminar series
  Interventions: Other: Wellness Seminar Series

INTERVENTIONS:
Other: Iyengar Yoga — The poses and breathing techniques to be used in this study are based on sequences developed by B.K.S. Iyengar for breast cancer survivors who suffer from fatigue. Women will start with simple versions of the poses and progress to more advanced versions over the course of the intervention.
  Other Names: Yoga
  Arms: 1
Other: Wellness Seminar Series — The Wellness Seminar Series consists of lectures on key topics, followed by group discussion. This series will focus entirely on cancer survivorship, including sessions on quality of life, side effects of cancer treatment, stress, nutrition and psychosocial issues.
  Other Names: Health education
  Arms: 2

SUMMARY:
This randomized controlled trial will compare the effectiveness of an Iyengar Yoga intervention to a Wellness Seminar health education lecture series, for improvements in energy, mood and biological functioning in breast cancer survivors with persistent, post-treatment fatigue. It is anticipated that the Iyengar Yoga intervention will be feasible and acceptable to breast cancer survivors with minimal side effects and that the Yoga intervention will be effective in improving fatigue and physical performance.

DETAILED DESCRIPTION:
Fatigue is the most common and distressing side effect of cancer treatment and persists beyond successful treatment completion in approximately 30% of breast cancer survivors, causing serious disruption in quality of life. Behavioral interventions incorporating physical activity or relaxation/stress management have demonstrated beneficial effects on cancer-related fatigue, although research in cancer survivors is limited. Mind-body interventions such as yoga are extremely popular among cancer patients and offer a promising alternative to traditional treatments. Research is needed to establish the feasibility and efficacy of these interventions in cancer populations, particularly those who are experiencing problems with fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early, resectable breast cancer (Stage I or II)
* Completed treatment with surgery, radiation, and/or chemotherapy between 6 months and 5 years previously
* No other cancer in last 5 years, including breast cancer recurrence
* Postmenopausal women
* Age 40 - 65
* Reporting persistent cancer-related fatigue

Exclusion Criteria:

* Evidence that fatigue is directly related to a medical or psychiatric disorder (e.g., untreated hypothyroidism, diabetes, anemia (defined as hematocrit < 24), chronic fatigue syndrome, current major depression, insomnia, sleep apnea, restless leg syndrome)
* Evidence that fatigue is related to other non-cancer related factors (e.g., shift work, recent change in activity or schedule)
* Physical problems or conditions that could make yoga unsafe (e.g., serious neck injuries, unstable joints; also severe cachexia, dizziness, bone pain, severe nausea, etc)
* Regular use of medications and/or behavioral therapies that would confound evaluation of IY, including regular participation in yoga classes
* Presence of medical conditions that involve the immune system and would confound immune evaluation (e.g., autoimmune disorder, inflammatory disease)
* Use of medications that might confound immune evaluation (e.g., regular use of corticosteroids, narcotics, opiates)
* Unable to commit to intervention schedule
* Body mass index greater than 30 kg/m2
* Regular tobacco (defined as daily or near daily) or alcohol use (defined as > 2 drinks/day)

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Fatigue | Measured at baseline, after the 12 week intervention and at 3 months post-intervention

SECONDARY OUTCOMES:
Secondary outcomes include depressed mood, sleep disturbance, pain, quality of life, and proinflammatory cytokine activity | Measured at baseline, after the 12 week intervention and at 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Julienne E Bower, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Cousins Center for PNI, Los Angeles, California, United States

REFERENCES:
- [Background] Bower JE, Woolery A, Sternlieb B, Garet D. Yoga for cancer patients and survivors. Cancer Control. 2005 Jul;12(3):165-71. doi: 10.1177/107327480501200304. PMID 16062164